CLINICAL TRIAL: NCT03068598
Title: Connected Sleep Recording Device for Suicidal Patients, Acceptability Study - Suicide Sleep Monitoring (Ssleem)
Brief Title: Suicide Sleep Monitoring (Ssleem)
Acronym: SSLEEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SSLEEM 29BRC16.0107
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2018-01

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: The subject will receive a watch connected to a smartphone, wear at night and objectively evaluate sleep in ecological conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sleep monitoring (Experimental): The sleep tracker and a smartphone will be given to the patient after discharge. The patient will recieve a brief training on how to use the PulseOn watch or the Suunto Spartan Ultra watch. Patient will be proposed to monitor his sleep during the five nights following the discharge.
  Interventions: Device: PulseOn watch/Suunto Spartan Ultra watch

INTERVENTIONS:
Device: PulseOn watch/Suunto Spartan Ultra watch — The Watch (PulseOn or Suunto Spartan Ultra) and a smartphone will be given to the patient after discharge. After a brief training on how to use the sleep tracker, patient will monitor his sleep with watch during the five nights following the discharge. All data will be transmitted directly to the smartphone. Each morning, the patient will complete a questionnaire to assess the quality of his sleep and on day 5, during a standart follow up visit, he will complete a questionnaire evaluating the acceptability of the sleep recording device.

SUMMARY:
Promising results have shown that interventions to reduce insomnia diminish suicidal ideation. A better understanding of the bidirectional mechanism between sleep disturbances and suicide behavior will allow the design of tailored interventions to prevent suicide attempts.

Significance of the proposed study for the field The aim of the present is to assess the feasibility and the acceptability of sleep tracking monitoring in a sample of suicide attempters. The investigator hypothesize that sleep monitoring using a connected object is feasable and acceptable by patients.

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged 18 or older,
* with suicide attempt or suicidal ideas history,
* able to understand the study,
* insured persons,
* having signed a consent form.

Exclusion Criteria:

* minor patient,
* patient whose clinical status is incompatible with informed consent,
* patient tattooed on both wrists
* patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Acceptability of the sleep recorder device in patients with previous history of suicide attempts | 5 days after discharge
  Score obtained at the scale evaluating acceptability of the sleep recorder device during the study exit interview 5 days after inclusion

SECONDARY OUTCOMES:
Link between the connected record and the data collected using a self-administered questionnaire evaluating qualitatively and quantitatively sleep. | 5 days after discharge
  Subjective evaluation of sleep by a validated questionnaire compared to the data of the sleep recording.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No